CLINICAL TRIAL: NCT03437265
Title: A Pharmacokinetic Study of PLENVU® in Healthy Subjects
Acronym: PKPU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NER1006-03/2016 (PKPU); 2017-003440-20 (EudraCT Number)
Record Dates: First submitted 2018-01-16; First posted 2018-02-19 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pharmacokinetic
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PLENVU powder for oral solution (Experimental): Dose 1: Oral administration of 1 sachet (115.96 g) PLENVU Dose 1, reconstituted with water and made up to 473 mL and 473 mL of additional water to be consumed; both to be consumed over a period of 60 min after the start of Dose 1.
  Dose 2: Oral administration of 2 sachets (101.91 g) comprising PLENVU Dose 2, reconstituted with water and made up to 473 mL and 473 mL of additional water to be consumed; both to be consumed over a period of 60 min after the start of Dose 2.
  Additional water was permitted ad libitum during and after each dose.
  Interventions: Drug: PLENVU powder for oral solution

INTERVENTIONS:
Drug: PLENVU powder for oral solution — PLENVU Dose 1 (1 sachet) and PLENVU Dose 2 (2 sachets)
  Other Names: NER1006

SUMMARY:
This study characterises the pharmacokinetic (PK) profile of the active ingredients of PLENVU (NER1006) and their related substances/metabolites. Subjects will receive PLENVU.

DETAILED DESCRIPTION:
PLENVU is a novel, low volume (1 L) PEG 3350 and ascorbate based bowel preparation that has been developed to provide whole bowel cleansing. Studies have shown that formulating the osmotically active agents sodium ascorbate/ascorbic acid (also known as vitamin C) and sodium sulfate in combination with PEG 3350 enable a reduction in the volume of the PEG-based lavage solution.

PLENVU has a dual formulation containing an initial majority PEG dose followed by a majority ascorbate dose to maximise the overall effectiveness. This novel formulation addresses the challenges faced by patients to comply with drinking higher volume, 2 and 3 L, preparations.

The purpose of this study is to determine if there is systemic exposure to components of the PLENVU formulation (PEG 3350, ascorbate and potential related substances/metabolites (oxalic acid, glycolic acid, ethylene glycol and diethylene glycol).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Age 18 to 30 years
3. BMI of 18.0 to 35.0 kg/m2
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Subjects who have received any Investigational Medicinal Product (IMP) in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study.
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. Females who are pregnant or lactating (all female subjects must have a negative urine pregnancy test at screening and admission).
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
10. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator at screening
11. Evidence of dehydration or abnormal electrolyte levels. Clinical evidence or suspicion of significant dehydration at admission/pre-dose.
12. History or evidence of any clinically relevant ECG abnormality and hypertension
13. Positive drugs of abuse test result
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
15. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or psychiatric disorder, as judged by the investigator
16. History or presence of organic or functional gastrointestinal conditions (e.g. chronic constipation, inflammatory bowel disease or irritable bowel syndrome)
17. Previous or current relevant abnormal gastrointestinal motility according to clinical judgement
18. History or presence of any clinically significant acute illness within 28 days prior to the first dose of IMP based on clinical judgement at screening or admission
19. History of any of the contraindications mentioned in the PLENVU Summary of Product Characteristics (SmPC)
20. Clinically relevant findings on physical examination based on investigator judgement
21. Donation or loss of greater than 500 mL of blood within the previous 8 weeks
22. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than hormonal contraception and occasional use of non-steroidal anti-inflammatory drugs [NSAIDs] and paracetamol) or herbal remedies in the 28 days before IMP administration Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
23. Use of laxatives and gastrointestinal motility altering drug in the last 3 months
24. Evidence of current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection
25. Subjects who are ordered to live in an institution on court or authority order
26. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, MRCS, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences (Quotient),, Ruddington, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Healthy adult subjects given PLENVU powder for oral solution: PLENVU Dose 1 (1 sachet) and PLENVU Dose 2 (2 sachets)
Period: Overall Study
Arm/Group | Overall Study
Started | 19
Completed | 13
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Population: Healthy adult subjects who recieved at least a partial dose of PLENVU
Groups:
- Overall Study: All subjects who received at least a partial dose of IMP
Arm/Group | Overall Study
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 25.0 [19 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19
BMI [Mean (Standard Deviation); unit: kg/m2] — Body mass index weight in kg/ height in m2
  kg/m2 | 24.85 (3.896)
Height [Mean (Standard Deviation); unit: cm] — Height in cm
  cm | 171.5 (10.92)
Weight [Mean (Standard Deviation); unit: kg] — Weight in kg
  kg | 73.82 (17.011)

OUTCOME MEASURES:

1. Primary Outcome: Tmax (PEG 3350, Baseline-corrected Glycolic Acid and Baseline-corrected Ascorbic Acid)
Description: Time of maximum observed concentration (of PEG3350, and glycolic acid and ascorbic acid corrected for baseline levels), calculated from individual plasma concentrations of the pharmacokinetic (PK) population.
Time Frame: Blood samples were taken pre-dose and up to 60 hours after start of Dose 1
Population: PK population 1: all evaluable subjects who had a minimum of 1 valid post-dose analytical result for PK parameter estimation and who satisfied the following criterion for at least 1 profile: no relevant protocol deviations which may have impacted the study objectives with respect to the PK endpoints.
Measure: Median (Full Range); unit: hours
Arm/Group | Overall Study
Number analyzed (Participants) | 13
hours
  PEG 3350 | 3.00 [1.97 to 4.03]
  Glycolic acid | 9.00 [4.00 to 36.07]
  Ascorbic acid | 5.00 [4.00 to 6.00]
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; PK parameters were estimated for each subject by non-compartmental analysis methods using Phoenix® WinNonlin® software (v8.0, Certara USA, Inc., USA). Summary statistics (n, mean, SD, CV%, median, minimum, maximum, geometric n, geometric mean (geometric SD) and geometric CV%) were presented

2. Primary Outcome: T1/2 (PEG 3350, Baseline-corrected Glycolic Acid and Baseline-corrected Ascorbic Acid)
Description: Apparent elimination half-life (of PEG3350, and glycolic acid and ascorbic acid corrected for baseline levels), calculated from individual plasma concentrations of the PK population.
Time Frame: Blood samples were taken pre-dose and up to 60 hours after start of Dose 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Overall Study
Number analyzed (Participants) | 13
hours
  PEG 3350 | 3.58 (14.3)
  Glycolic acid | 4.63 (0)
  Ascorbic acid | 11.62 (270)
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Cmax (PEG 3350, Baseline-corrected Glycolic Acid and Baseline-corrected Ascorbic Acid)
Description: The mean maximum observed concentration (of PEG3350, and glycolic acid and ascorbic acid corrected for baseline levels), calculated from individual plasma concentrations of the PK population.
Time Frame: Blood samples were taken pre-dose and up to 60 hours after start of Dose 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Overall Study
Number analyzed (Participants) | 13
ng/mL
  PEG 3350 | 1010 (42.5)
  Glycolic acid | 528 (113.0)
  Ascorbic Acid (μg/mL) | 59.1 (26.1)
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Area Under the Curve From 0 Time to 24 h Post-dose (AUC[0-24]) (PEG 3350, Baseline-corrected Glycolic Acid and Baseline-corrected Ascorbic Acid)
Description: Area under the curve from 0 time to 24 h post-dose (of PEG3350, and glycolic acid and ascorbic acid corrected for baseline levels), calculated from individual plasma concentrations of the PK population.
Time Frame: Blood samples were taken pre-dose and up to 60 hours after start of Dose 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Overall Study
Number analyzed (Participants) | 13
ng.h/mL
  PEG 3350 | 7220 (31.7)
  Glycolic acid | 3820 (53.1)
  Ascorbic acid (μg.h/mL) | 359 (17.3)
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; [other analysis details as in outcome 1, analysis 1]

5. Primary Outcome: AUC(0-last) (PEG 3350, Baseline-corrected Glycolic Acid and Baseline-corrected Ascorbic Acid)
Description: Area under the curve from 0 time to the last measurable concentration (of PEG3350, and glycolic acid and ascorbic acid corrected for baseline levels), calculated from individual plasma concentrations of the PK population.
Time Frame: Blood samples were taken pre-dose and up to 60 hours after start of Dose 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Overall Study
Number analyzed (Participants) | 13
ng.h/mL
  PEG 3350 | 7140 (32.2)
  Glycolic acid | 9020 (51.5)
  Ascorbic acid (μg.h/mL) | 437 (24.0)
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; [other analysis details as in outcome 1, analysis 1]

6. Primary Outcome: AUC(0-inf) (PEG 3350, Baseline-corrected Glycolic Acid and Baseline-corrected Ascorbic Acid)
Description: Area under the curve from 0 time extrapolated to infinity (of PEG3350, and glycolic acid and ascorbic acid corrected for baseline levels), calculated from individual plasma concentrations of the PK population.
Time Frame: Blood samples were taken pre-dose and up to 60 hours after start of Dose 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Overall Study
Number analyzed (Participants) | 13
ng.h/mL
  PEG 3350 | 7340 (31.1)
  Gycolic acid | 6900 (0)
  Ascorbic acid (μg.h/mL) | 397 (23.9)
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; PK parameters were estimated for each subject by non-compartmental analysis methods using Phoenix® WinNonlin® software (v8.0, Certara USA, Inc., USA). Summary statistics (n, mean, SD, CV%, median, minimum, maximum, geometric n, geometric mean (geometric SD) and geometric CV%) were presented. The Geometric CV for glycolic acid was Not Calculated (appears as 0%)

7. Secondary Outcome: Timing and Number of Bowel Movements
Description: Pharmacodynamic outcome. The time of each bowel movement will be recorded for each subject, and the number of bowel movements after each dose per subject will be derived.
Time Frame: Start of dose 1 to 60 hours
Population: Pharmacodynamic (PD) analysis set: subjects who received both doses and had sufficient PD data for at least 1 time point
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  0-6 hours: 0 bowel movements | 0
  0-6 hours: 1 bowel movement | 0
  0-6 hours: 2 bowel movements | 1
  0-6 hours: 3 bowel movements | 0
  0-6 hours: 4 bowel movements | 1
  0-6 hours: 5 bowel movements | 2
  0-6 hours: 6 bowel movements | 1
  0-6 hours: 7 bowel movements | 4
  0-6 hours: 8 bowel movements | 0
  0-6 hours: 9 bowel movements | 1
  0-6 hours: ≥10 bowel movements | 3
  6 - 12 hours: 0 bowel movements | 1
  6 - 12 hours: 1 bowel movement | 4
  6 - 12 hours: 2 bowel movements | 4
  6 - 12 hours: 3 bowel movements | 4
  6 - 12 hours: 4 bowel movements | 0
  6 - 12 hours: 5 bowel movements | 0
  6 - 12 hours: 6 bowel movements | 0
  6 - 12 hours: 7 bowel movements | 0
  6 - 12 hours: 8 bowel movements | 0
  6 - 12 hours: 9 bowel movements | 0
  6 - 12 hours: ≥10 bowel movements | 0
  12 - 24 hours: 0 bowel movements | 10
  12 - 24 hours: 1 bowel movement | 3
  12 - 24 hours: 2 bowel movements | 0
  12 - 24 hours: 3 bowel movements | 0
  12 - 24 hours: 4 bowel movements | 0
  12 - 24 hours: 5 bowel movements | 0
  12 - 24 hours: 6 bowel movements | 0
  12 - 24 hours: 7 bowel movements | 0
  12 - 24 hours: 8 bowel movements | 0
  12 - 24 hours: 9 bowel movements | 0
  12 - 24 hours: ≥10 bowel movements | 0
  24 - 48 hours: 0 bowel movements | 10
  24 - 48 hours: 1 bowel movement | 3
  24 - 48 hours: 2 bowel movements | 0
  24 - 48 hours: 3 bowel movements | 0
  24 - 48 hours: 4 bowel movements | 0
  24 - 48 hours: 5 bowel movements | 0
  24 - 48 hours: 6 bowel movements | 0
  24 - 48 hours: 7 bowel movements | 0
  24 - 48 hours: 8 bowel movements | 0
  24 - 48 hours: 9 bowel movements | 0
  24 - 48 hours: ≥10 bowel movements | 0
  48 - 60 hours: 0 bowel movements | 10
  48 - 60 hours: 1 bowel movement | 3
  48 - 60 hours: 2 bowel movements | 0
  48 - 60 hours: 3 bowel movements | 0
  48 - 60 hours: 4 bowel movements | 0
  48 - 60 hours: 5 bowel movements | 0
  48 - 60 hours: 6 bowel movements | 0
  48 - 60 hours: 7 bowel movements | 0
  48 - 60 hours: 8 bowel movements | 0
  48 - 60 hours: 9 bowel movements | 0
  48 - 60 hours: ≥10 bowel movements | 0
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; Summary of the number of bowel movements per time period for the PD analysis set

8. Secondary Outcome: Time to Achieve Clear Effluent
Description: Pharmacodynamic outcome. Scoring was according to a 4-point scale (adapted from the stool characteristics rating tool described by Hsu et al, Adv Dig Med. 2016; 3 (3):144-147).
  A. Clear contents (may be coloured but able to visualise the bottom of the toilet bowl) B. Turbid contents C. Opaque contents (dark and murky) D. Any solid/semi-solid faecal material (irrespective of size) in the toilet bowl
Time Frame: Start of dose 1 to 60 hours
Population: PD (pharmacodynamic) analysis set: subjects who received both doses and had sufficient PD data for at least 1 time point
Measure: Mean (Full Range); unit: minutes
Arm/Group | Overall Study
Number analyzed (Participants) | 13
minutes
  Time to clear effluent (A): number analyzed (Participants) | 10
  Time to clear effluent (A) | 226.0 [98 to 310]
  Time to turbid contents (B) | 165.5 [58 to 410]
Statistical Analysis 1: Comparison: Overall Study; Test type: Other; The time (in minutes) to achieve clear effluent/time to turbid contents is presented for the PD analysis set

ADVERSE EVENTS:
Time Frame: Screening (Day -28 to -2) to post study follow-up (Day 6 to 8)
Description: Adverse Events were recorded from the time of providing written informed consent until discharge from the study at the follow-up visit/call. During each study visit, subjects were questioned directly regarding the occurrence of any adverse medical event according to the schedule in the clinical database.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=19)
Diarrhoea (Gastrointestinal disorders) | 19 (19)
Nausea (Gastrointestinal disorders) | 8 (8)
Proctalgia (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Feeling hot (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
In addition to PEG 3350, glycolic acid and ascorbic acid, PK parameters were to be determined for oxalic acid, ethylene glycol and diethylene glycol. However, this was not done, as no quantifiable concentrations of oxalic acid (LLOQ <10.0 μg/mL), diethylene glycol (LLOQ <2.50 μg/mL), or ethylene glycol (LLOQ <2.50 μg/mL) were observed.

Diarrhoea was expected as it is the intended pharmacodynamic effect of PLENVU bowel preparation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement between Norgine and Quotient Sciences states that Quotient have no publication rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03437265/Prot_SAP_001.pdf